CLINICAL TRIAL: NCT01533077
Title: Pharmacokinetic Interaction Between BIA 9-1067 and Standard-release Levodopa/Carbidopa in Healthy Subjects
Brief Title: Pharmacokinetic Interaction Between BIA 9-1067 and Standard-release Levodopa/Carbidopa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-117
Record Dates: First submitted 2012-01-24; First posted 2012-02-15 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; carbidopa, levodopa drug combination; Levodopa; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Period 1: BIA 9-1067 50 mg Period 2: Sinemet® 100/25 1 h after the BIA 9-1067 50 mg Period 3: BIA 9-1067 50 mg + Sinemet® 100/25 Period 4: Sinemet® 100/25
  Interventions: Drug: BIA 9-1067; Drug: Sinemet® 100/25 mg
- Group 2 (Experimental): Period 1: Sinemet® 100/25 Period 2: BIA 9-1067 50 mg Period 3: Sinemet® 100/25 1 h after the BIA 9-1067 50 mg Period 4: BIA 9-1067 50 mg + Sinemet® 100/25
  Interventions: Drug: BIA 9-1067; Drug: Sinemet® 100/25 mg
- Group 3 (Experimental): Period 1: BIA 9-1067 50 mg + Sinemet® 100/25 Period 2: Sinemet® 100/25 Period 3: BIA 9-1067 50 mg Period 4: Sinemet® 100/25 1 h after the BIA 9-1067 50 mg
  Interventions: Drug: BIA 9-1067; Drug: Sinemet® 100/25 mg
- Group 4 (Experimental): Period 1: Sinemet® 100/25 1 h after the BIA 9-1067 50 mg Period 2: BIA 9-1067 50 mg + Sinemet® 100/25 Period 3: Sinemet® 100/25 Period 4: BIA 9-1067 50 mg
  Interventions: Drug: BIA 9-1067; Drug: Sinemet® 100/25 mg

INTERVENTIONS:
Drug: BIA 9-1067 — 50 mg of BIA 9-1067 (single-dose)
  Other Names: OPC, Opicapone
Drug: Sinemet® 100/25 mg — immediate-release levodopa/carbidopa 100/25 (single-dose).
  Other Names: levodopa 100 mg /carbidopa 25 mg

SUMMARY:
To investigate the pharmacokinetics of levodopa when administered concomitantly with BIA 9-1067 or 1 hour after.

DETAILED DESCRIPTION:
Single-centre, open-label, randomized, gender-balanced, crossover study with four consecutive single-dose treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period and willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer prior to participation in the study.
* Male or female volunteers.
* Volunteers of at least 18 years of age but not older than 45 years.
* Volunteers with body mass index (BMI) greater than or equal to 19 and below 30 kg/m2.
* Volunteers who were healthy as determined by pre-study (at screening) medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Volunteers who had clinical laboratory test results judged clinically acceptable (within the laboratory's stated normal range; if not within this range, they must had been without any clinical significance) at screening and admission to first treatment period.
* Volunteers who had negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibodies (HCV Ab), and Human immunodeficiency viruses -1 and -2 antibodies (HIV-1 and HIV-2 Ab) at screening.
* Volunteers who had negative screen of ethyl alcohol and drugs of abuse at screening.
* Volunteers who were non- or ex-smokers. For the purpose of this study, an ex-smoker is defined as someone who completely stopped smoking for at least 3 months before day 1 of this study.
* Due to unknown risks and potential harm to the unborn fetus, sexually active men or women must have agreed to use a medically acceptable form of contraception throughout the study.
* If female of childbearing potential, she had a negative HCG beta serum pregnancy test at screening and admission to each treatment period
* The informed consent form must have been signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

* Volunteers who did not conform to the above inclusion criteria, or in case of
* Volunteers who had a clinically relevant surgical history.
* Volunteers who had a clinically relevant family history.
* Volunteers who had a history of relevant atopy.
* Volunteers who had a significant infection or known inflammatory process at screening or admission to the treatment period.
* Volunteers who had acute gastrointestinal symptoms at the time of screening or admission to the treatment period (e.g., nausea, vomiting, diarrhoea, heartburn).
* Volunteers who were vegetarians, vegans or have medical dietary restrictions.
* Volunteers who could not communicate reliably with the investigator.
* Volunteers who were unlikely to co-operate with the requirements of the study.
* History of hypersensitivity to BIA 9-1067, tolcapone, entacapone, levodopa, benserazide or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability.
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, lymphatic, musculoskeletal, genitourinary, endocrine, immunologic, dermatologic or connective tissue disease.
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases.
* Presence of significant heart disease or disorder according to ECG.
* Presence of suspicious undiagnosed skin lesions or a history of melanoma.
* Previous history of Neuroleptic Malignant Syndrome (NMS) and/or nontraumatic rhabdomyolysis.
* History of significant glaucoma.
* Used of prescription medications including monoamine oxidase (MAO) inhibitors within 28 days before day 1 of the study.
* Used of over-the-counter (OTC) products within 7 days before day 1 of the study.
* Maintenance therapy with any drug, or significant history of drug dependency (drug abuse) or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic).
* Any clinically significant illness in the previous 28 days before day 1 of this study.
* Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study.
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician.
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
* Positive urine screening of ethyl alcohol or drugs of abuse at admission to the treatment period.
* Any history of tuberculosis and/or prophylaxis for tuberculosis.
* Positive results to HIV, HBsAg or anti-HCV tests.
* Participation in any previous clinical study with BIA 9-1067 within 84 days before day 1 of the study.
* Females who were pregnant according to a positive serum pregnancy test or were lactating.
* Females of childbearing potential who refused to use an acceptable contraceptive regimen throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 5 | 5 | 4 | 4
BIA 9-1067 50 mg | 5 | 5 | 4 | 4
Sinemet® 100/25 | 4 | 5 | 4 | 4
BIA 9-1067 50 mg + Sinemet® 100/25 | 4 | 4 | 4 | 4
Sinemet® 100/25 1 h After the BIA 9-1067 | 5 | 5 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 4 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 3 | 3 | 2 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (L-DOPA)
Description: Mean pharmacokinetic parameters of L-beta-3,4-dihydroxyphenylalanine (levodopa) (L-DOPA)
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: According to the protocol, the "pharmacokinetic population" should include all subjects who had valid data for all treatment periods. In this study, 18 subjects completed 2 treatment periods, 17 subjects completed 3 treatment periods and 16 subjects completed all 4 treatment periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sinemet® 100/25 mg: Levodopa 100 mg Carbidopa 25 mg
- BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h: BIA 9-1067 50 mg + Sinemet® 100/25 mg separated 1 h BIA 9-1067 Levodopa 100 mg Carbidopa 25 mg
- BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly: BIA 9-1067 50 mg + Sinemet® 100/25 mg concomitantly BIA 9-1067 Levodopa 100 mg Carbidopa 25 mg
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng/mL | 1070 (328) | 1105 (363) | 1198 (294)

2. Primary Outcome: Tmax - Time of Occurrence of Cmax Maximum Observed Plasma Concentration (L-DOPA)
Description: Pharmacokinetic parameters of L-beta-3,4-dihydroxyphenylalanine (levodopa) (L-DOPA). For tmax = time to Cmax values are presented as median with range values.
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
hours | 1.0 [0.5 to 2.0] | 1.0 [0.5 to 4.0] | 0.5 [0.5 to 1.0]

3. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point (L-DOPA)
Description: Mean pharmacokinetic parameters of L-beta-3,4-dihydroxyphenylalanine (levodopa) (L-DOPA)
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 2289 (729) | 2611 (916) | 2459 (825)

4. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (L-DOPA)
Description: Mean pharmacokinetic parameters of L-beta-3,4-dihydroxyphenylalanine (levodopa) (L-DOPA)
Time Frame: pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 2397 (741) | 2730 (913) | 2603 (836)

5. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (3-OMD)
Description: Mean pharmacokinetic parameters of 3-O-methyl-levodopa (3-OMD)
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng/mL | 490 (175) | 336 (127) | 401 (141)

6. Primary Outcome: Tmax - Time to Occurrence of Cmax (3-OMD)
Description: Pharmacokinetic parameters of 3-O-methyl-levodopa (3-OMD). For tmax = time to Cmax values are presented as median with range values.
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
hours | 6.00 [4.00 to 6.00] | 5.00 [4.00 to 8.00] | 5.00 [3.00 to 8.00]

7. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point (3-OMD)
Description: Mean pharmacokinetic parameters of 3-O-methyl-levodopa (3-OMD)
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 10296 (3151) | 6940 (2504) | 8149 (2809)

8. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (3-OMD)
Description: Mean pharmacokinetic parameters of 3-O-methyl-levodopa (3-OMD)
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 11193 (3187) | 7730 (2578) | 89962 (2803)

9. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (Carbidopa)
Description: Mean pharmacokinetic parameters of carbidopa
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng/mL | 134 (56.2) | 136 (62.0) | 142 (71.3)

10. Primary Outcome: Tmax - Time to Occurrence of Cmax (Carbidopa)
Description: Pharmacokinetic parameters of carbidopa. For tmax = time to Cmax values are presented as median with range values.
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
hours | 3.00 [1.50 to 4.00] | 3.00 [1.00 to 4.00] | 3.00 [1.00 to 4.00]

11. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point (Carbidopa)
Description: Mean pharmacokinetic parameters of carbidopa
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 656 (226) | 670 (253) | 732 (335)

12. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (Carbidopa)
Description: Pharmacokinetic parameters of carbidopa. For tmax = time to Cmax values are presented as median with range values.
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sinemet® 100/25 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 18 | 16
ng.h/mL | 668 (224) | 683 (253) | 745 (337)

13. Primary Outcome: Cmax - Maximum Observed Plasma Concentration (BIA 9-1067)
Description: Mean pharmacokinetic parameters of BIA 9-1067
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 50 mg: BIA 9-1067 50 mg
Arm/Group | BIA 9-1067 50 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 18 | 18 | 16
ng/mL | 648 (264) | 625 (346) | 628 (295)

14. Primary Outcome: Tmax - Time to Occurrence of Cmax (BIA 9-1067)
Description: Pharmacokinetic parameters of BIA 9-1067. For tmax = time to Cmax values are presented as median with range values.
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 50 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 18 | 18 | 16
hours | 2.50 [1.00 to 6.00] | 3.50 [0.50 to 6.00] | 4.00 [2.00 to 6.00]

15. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve to Last Measurable Time Point (BIA 9-1067)
Description: Mean pharmacokinetic parameters of BIA 9-1067
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 50 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 18 | 18 | 16
ng.h/mL | 2094 (904) | 2130 (1248) | 2245 (1171)

16. Primary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity (BIA 9-1067)
Description: Mean pharmacokinetic parameters of BIA 9-1067
Time Frame: Pre-dose, ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 h after dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 50 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly
Number analyzed (Participants) | 17 | 15 | 11
ng.h/mL | 2165 (913) | 2360 (1281) | 2678 (1334)

ADVERSE EVENTS:
Groups:
- BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h: BIA 9-1067 50 mg + Sinemet® 100/25 mg separated 1 h.
- BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly: BIA 9-1067 50 mg + Sinemet® 100/25 mg concomitantly.
- Sinemet® 100/25 mg: Sinemet® 100/25 mg.
Arm/Group | BIA 9-1067 50 mg | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly | Sinemet® 100/25 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/18 | 10/18 | 8/16 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 50 mg (N=18) | BIA 9-1067 50 mg + Sinemet® 100/25 mg Separated 1 h (N=18) | BIA 9-1067 50 mg + Sinemet® 100/25 mg Concomitantly (N=16) | Sinemet® 100/25 mg (N=17)
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure systolic decreased (Investigations) | 0 | 0 | 0 | 1
Blood pressure systolic increased (Investigations) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 4 | 4
Somnolence (Nervous system disorders) | 6 | 4 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other